CLINICAL TRIAL: NCT03215654
Title: "EspaiJove.Net"- a School-based Intervention Program to Promote Mental Health and Eradicating Stigma in Adolescent Population: a Randomised Controlled Trial
Brief Title: "EspaiJove.Net"- a School-based Intervention Program to Promote Mental Health in Adolescent Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Higiene Mental Les Corts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PI15/01613
Record Dates: First submitted 2017-07-04; First posted 2017-07-12 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Mental Health; Stigma, Social
Keywords: mental health; promotion; prevention; adolescence; school programs; intervention
MeSH Terms: conditions — Psychological Well-Being; Social Stigma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sensitization Program (SP) (Experimental): Include the concepts of mental health and mental disorder, healthy and risky behaviors of mental health, and use of health services. Duration 1 hour.
  Interventions: Other: "EspaiJove.net" mental health literacy program
- Mental Health Literacy Program (MHL) (Experimental): MHL module contents are: 1) Our emotions. Definitions of mental health and mental disorders. Mental health multidisciplinary team network; 2) Healthy and risky behaviors of mental health; 3) Social skills and antisocial behavior, bullying and cyberbullying; 4) Anxiety, depression, self-harm, and suicidal behaviors; 5) Eating and behavioral disorders; 6) Substance abuse (alcohol and cannabis), an psychotic disorder. Duration 6 hours.
  Interventions: Other: "EspaiJove.net" mental health literacy program
- MHL more Stigma Reduction (ER) (Experimental): Includes the six teaching units of MHL and a first contact presentation with lived experience of any mental disorder, who will be delivered by a voluntary member of Activament Catalunya Associació (http://www.activament.org/es), a non-profit group specialized in reducing stigma. Duration 7 hours.
  Interventions: Other: "EspaiJove.net" mental health literacy program
- Control group (No Intervention): Control group will be a waiting list condition and they will receive the full program of 7h at the next year of academic course

INTERVENTIONS:
Other: "EspaiJove.net" mental health literacy program — The "EspaiJove.net: a space for mental health" (EspaiJove.net) project is a MHL program which aims the promotion of mental health, the prevention of mental disorders, the facilitation of help-seeking behaviors and the eradication of stigma among secoundary students into the Spanish context.
  Arms: MHL more Stigma Reduction (ER); Mental Health Literacy Program (MHL); Sensitization Program (SP)

SUMMARY:
Objective: To evaluate the efficacy of 3 sensitivity and mental health literacy programs for young students in the increase of mental health knowledge, to help seeking and reducing the stigma in order to prevent mental disorders and to reduce symptoms.

Design: Multicenter randomized clinical trial school-based during 12 months follow up. Setting: Educational centers of secondary education (E.S.O) (public or private) of Barcelona. Subjects: 408 students between 13 and 18 years old who attend 3rt ESO in 8 randomized schools of Barcelona.

Interventions: 3 intervention groups of ascending intensity: 1) Sensitivity Program Mental Health (SP)(1h); 2) Mental Health Literacy Program (MHLP) (6h); 3) MHLP more Stigma Reduction (ER) ( MHLP+RE)(7h).Control group: waiting List.

Measures of results:1) Mental Health Literacy; 2) Stigma associated with mental health; 3) Mental Symptoms and Positive Mental Health (SDQ); 4) Bullying and Ciberbullying; 5) Quality of life (E-5D); 6) Intent to change; 7) Help Seeking (AHSQ); 8) Use of Health Services and Treatment and 9) Satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents students who are currently attending the 3rd grade of E.S.O (corresponding to 9th grade in U.S.) in Barcelona, Spain;
* Sign the informed consent

Exclusion Criteria:

* Attending any special education school;
* Students with special educational needs who attend any school;
* Not understanding Spanish and Catalan language.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 432 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Change in the Mental Health knowledge | Change from Baseline to 2 weeks after the intervention, 6 months and 12 months after the intervention.
  This questionnaire is divided by two sections: (a) an identification list of mental disorders from a list of several diseases; (b) 20 questions with 4 possible answer choices which only one is correct.
Change in the Scaling Community Attitudes toward the Mentally Ill (CAMI). | Change from Baseline to 2 weeks after the intervention, 6 months and 12 months after the intervention.
  Behaviour and Attitudes towards Mental health ( stigma)

SECONDARY OUTCOMES:
Change in the Mental health symptoms and emotional well-being | Change from Baseline to 2 weeks after the intervention, 6 months and 12 months after the intervention.
  The Strengths and Difficulties Scale (SDQ) will assess mental health symptoms and emotional well-being.
Change in the Bullying and Cyberbullying questionnaire | Change from Baseline to 2 weeks after the intervention, 6 months and 12 months after the intervention.
  We developed four yes/no questions to ask whether he/she has been a victim or perpetrator of a bullying and/or a cyberbullying experience.
Change in the Quality of life | Change from Baseline to 2 weeks after the intervention, 6 months and 12 months after the intervention.
  We will use a Spanish validated version of the EuroQol 5D-5L questionnaire (EQ-5D-5L)
Change in the Intentions to Change | Change from Baseline to 2 weeks after the intervention, 6 months and 12 months after the intervention.
  We will use the adapted Spanish version of the States of Change Scale (SCS). This is based on the Transtheoretical Change Model developed by J. Prochaska and C. DiClemente to assess the degree intention, disposition or attitude towards change.
Change in the Help-seeking | Change from Baseline to 6 months and 12 months after the intervention.
  We selected and adapted the first item from the Spanish version of the General Help-Seeking Questionnaire (GHSQ) for measuring help-seeking behaviour in adolescents.
Change in the Use of Health Services and Treatment | Change from Baseline to 6 months and 12 months after the intervention.
  We developed a 8- ítems questionnaire to evaluate the use of health services and treatment
Health Benefits Questionnaire | Baseline
  We developed a 17-items questionnaire to evaluate family, academic and general health benefits.
Acceptability and satisfaction of the intervention | 2 weeks after the intervention
  We developed a short questionnaire for assessing acceptability and satisfaction to measure the degree of receptivity of the people to the interventions proposed.
Change in the Reported and Intended Behaviour Scale (RIBS) | Change from Baseline to 2 weeks after the intervention, 6 months and 12 months after the intervention.
  Behaviour and Attitudes towards Mental health ( stigma)

CONTACTS AND LOCATIONS:
Overall Officials: Lluis Lalucat, Principal Investigator — Centre Higiene Mental Les Corts
Locations (2):
- Spain (2):
  - Centre Higiene Mental Les Corts, Barcelona
  - Rocio Casañas, Barcelona

REFERENCES:
- [Derived] Casanas R, Castellvi P, Gil JJ, Torres-Torres M, Baron J, Teixido M, Sampietro HM, Diez M, Fernandez R, Sorli R, Sinol P, Jurado F, Carreras-Salvador R, Vazquez D, Gonzalez S, Martin MIF, Raya-Tena A, Alvarez R, Amado-Rodriguez I, Lopez LMM, Alonso J, Lalucat-Jo L. The effectiveness of a "EspaiJove.net"- a school-based intervention programme in increasing mental health knowledge, help seeking and reducing stigma attitudes in the adolescent population: a cluster randomised controlled trial. BMC Public Health. 2022 Dec 24;22(1):2425. doi: 10.1186/s12889-022-14558-y. PMID 36566192
- [Derived] Casanas R, Arfuch VM, Castellvi P, Gil JJ, Torres M, Pujol A, Castells G, Teixido M, San-Emeterio MT, Sampietro HM, Caussa A, Alonso J, Lalucat-Jo L. "EspaiJove.net"- a school-based intervention programme to promote mental health and eradicate stigma in the adolescent population: study protocol for a cluster randomised controlled trial. BMC Public Health. 2018 Jul 31;18(1):939. doi: 10.1186/s12889-018-5855-1. PMID 30064404
- See also: Related Info — http://www.espaijove.net/index.php?lang=es